CLINICAL TRIAL: NCT04452474
Title: A Multicenter, Randomized, Double-blind, Adaptive, Placebo-controlled Study of the Efficacy and Safety of a Single Administration of Olokizumab vs. Placebo in Addition to Standard Treatment in Patients With Severe SARS-CoV-2 Infection (COVID-19)
Brief Title: Study of the Efficacy and Safety of a Single Administration of Olokizumab vs. Placebo in Addition to Standard Treatment in Patients With Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection (COVID-19).
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: R-Pharm (Industry)
Collaborators: Cromos Pharma LLC (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04041080
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; 2019-nCoV; 2019 novel coronavirus; Respiratory disease; lung disease; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Respiration Disorders; Lung Diseases; Coronavirus Infections | interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Olokizumab 64 mg (Experimental): Subject randomized to receive subcutaneous single injection of 0,4 ml solution of Olokizumab on Day 1, in addition to standard therapy
  Interventions: Drug: Olokizumab 64 mg
- Placebo (Placebo Comparator): Subject randomized to receive subcutaneous single injection of 0,4 ml solution of Placebo on Day 1, in addition to standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olokizumab 64 mg — solution for subcutaneous administration 160 mg/mL
  Arms: Olokizumab 64 mg
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution for Injection), in the market package
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of a single dose of OKZ (64 mg) vs placebo in addition to standard therapy in patients with severe SARS-CoV-2 infection (COVID-19) at Day 29.

DETAILED DESCRIPTION:
1. Pilot phase: the first 100 patients will be randomized in two groups to receive OKZ or placebo (50 patients per group). Early futility analysis will be performed based on the results obtained in the pilot period after 100th patient completed Visit 29. Enrollment will be paused after randomization of 100th patient, then interim analysis will be performed when all 100 patients complete Visit Day 29 or discontinue the study.Based on results of the pilot phase analysis the study could be stopped.
2. Pivotal phase: inclusion of patients until targeted sample size is reached and performing final safety and efficacy analysis.

Maximum expected study duration for each patient is 62 days, including 2 days of screening, 1 day of study drug administration, and 59 days of follow-up.

The study will include following periods:

1. Screening period lasting up to 48 hours prior to Day 1. After signing the informed consent by the patient or the legally acceptable representative or when prior consent of the patient is not possible, and the subject's legally acceptable representative is not available, after obtaining documented approval/favorable opinion for individual cases by the Institutional Review Board / Independent Ethic Committee (IRB/IEC), investigator will assess the subject's eligibility for the study.
2. Treatment period lasting from the beginning of Day 1 visit to 23:59 of the Day 1.

   Eligible patients will be randomized to one of two treatment groups to receive a single subcutaneous injection - OKZ 64 mg or placebo in addition to standard COVID-19 therapy according to institutional guidelines;
3. Follow-up period lasting from 00:00 of the Day 2 to 23:59 of the Day 60. If the patient is discharged earlier than Day 15, at Days 15 and 29 5-point clinical status scale will be assessed at the study site visit or by phone interview. If the patient is discharged after Day 15, but earlier than Day 29, at Day 29 5-point clinical status scale will be assessed at the study site visit or by phone interview. The end of study is Day 60, when 5-point clinical status scale will be assessed by phone interview.

Up to 376 randomized patients (full sample size) will be included in the study according to preliminary estimation.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnosis (confirmation of the presence of SARS-CoV-2 virus by rt-PCR) OR sample collection for SARS-CoV-2 virus rt-PCR if the results of SARS-CoV-2 virus rt-PCR are not available yet.
* Dated informed consent for participation in this study signed by the patient, or by the legally acceptable representative or when prior consent of the patient is not possible, and the subject's legally acceptable representative is not available, documented approval / favorable opinion by the IRB/IEC.
* SpO2 ≤93% (room air) or respiratory rate greater than 30/min (room air) or oxygenation index PaO2/FiO2 ≤300 mmHg (or SpO2/FiO2 ≤315 in the case PaO2/FiO2 assessment is not available (supplementary oxygen)
* Computed tomography findings: features consistent with bilateral COVID-19 viral pneumonia and no alternative explanation for these findings.

Exclusion Criteria:

* Presence of any of the following laboratory abnormalities:

absolute neutrophil counts <0,5 х 10^9/L white blood cell count < 2 х 10^9/L, platelet count < 50 х 10^9/L, Alanine aminotransferase (АLT) and/or Aspartate aminotransferase (AST) ≥3,0 х Upper Limit of Normal (ULN)

* Kidney injury with creatinine clearance <30 mL/min.
* Hypersensitivity to OKZ, and/or its components.
* Septic shock (need for vasopressors to maintain mean arterial pressure ≥ 65 mm Hg and lactate ≥2 mmol / L in the absence of hypovolemia).
* Estimated survival of less than 24 hours regardless of treatment.
* History of perforation of the gastrointestinal tract, history of diverticulitis.
* Recent (less than 5 half-lives), current or planned during the current study period use of immunosuppressive drugs:
* biologics (except OKZ) with immunosuppressive effect, including, but not limited to: Interleukin-1 (IL-1) inhibitors (anakinra, rilonacept, canakinumab), IL-6 inhibitors (tocilizumab, sarilumab, siltuximab, etc.), IL-17A inhibitors (seсukinumab, etc.), Tumor Necrosis Factor-alpha (TNF-alpha) inhibitors (infliximab, adalimumab, etanercept, etc.), anti-B-cells therapy, etc.;.
* other immunosuppressive drugs (excluding methotrexate in dose up to 25 mg/week), including but not limited to:

  1. Glucocorticoids in high doses (> 1 mg / kg equivalent of methylprednisolone) orally and parenterally;
  2. JAK inhibitors; etc.
* Concurrent participation in another clinical trial during 30 days before screening.
* Pregnancy or lactation.
* A history of active tuberculosis, or active tuberculosis suspected by the Investigator.
* Administration of plasma from COVID-19 reconvalescent donors for 4 weeks prior to the patient's inclusion in the study and/or planned administration during the study
* Patients who deteriorated into Category 4 of the 5-point clinical status scale within more than the last 24 hours.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-11-16 (Estimated); Study Completion 2021-01-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects achieving a change in their clinical status defined as improvement for at least 2 categories of the 5-points clinical status scale relative to baseline or in the "Not hospitalized" category | at Day 29
  Difference between OKZ and placebo groups in the percentage of subjects with an improvement of at least 2 categories of the 5-points clinical status scale relative to baseline or in the "Not hospitalized" category. The points of the scale are: 1. Not hospitalized; 2.Hospitalized, not requiring supplemental oxygen; 3.Hospitalized, supplemental oxygen, spontaneous breathing;4. Hospitalized, mechanical ventilation (invasive/non-invasive) or extracorporeal membrane oxygenation (ECMO); 5. Death

SECONDARY OUTCOMES:
Subjects' clinical status distribution based on 5-point clinical status scale during the study | from Day 2 tо Day 15, Day 29, Day 60
  Subjects' clinical status distribution based on 5-point clinical status scale during the study
28-day case fatality rates | from Day 1 to Day 29
  28-day case fatality rates

OTHER OUTCOMES:
Case fatality rates during the intensive care unit (ICU) stay, at Days 7, 15, and 60 | from Day 1 to Day 60
  Case fatality rates during the intensive care unit (ICU) stay at Days 7, 15, and 60
Duration of oxygen support | From Day 1 to Day 60
  Duration of oxygen support (if applicable)
The time period until SpO2 ≥ 94% at ambient air during 2 consequence days is reached | from Day 2 to Day 60
  The time period until SpO2 ≥ 94% at ambient air during 2 consequence days is reached
Changes of oxygenation index PaO2/FiO2 from baseline | from Day 2 to Day 60
  Changes of oxygenation index PaO2/FiO2 from baseline (if applicable)
Duration of oxygen support (if applicable) | from Day 1 to Day 60
  Duration of oxygen support (if applicable), in days
Duration of mechanical ventilation and/or ECMO (if applicable) | from Day 1 to Day 60
  Duration of mechanical ventilation and/or ECMO (if applicable), in days
Duration of ICU stay (if applicable) | from Day 1 to Day 60
  Duration of ICU stay (if applicable)
Changes from baseline of COVID-19 cytokine storm surrogate marker: white blood count | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker: white blood count
Changes from baseline of COVID-19 cytokine storm surrogate marker: lymphocyte count | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker: lymphocyte counts
Changes from baseline of COVID-19 cytokine storm surrogate marker: neutrophils count | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker: neutrophils count
Changes from baseline of COVID-19 cytokine storm surrogate marker: C-reactive protein (CRP) | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker: C-reactive protein (CRP)
Changes from baseline of COVID-19 cytokine storm surrogate marker: ferritin | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker: ferritin
Changes from baseline of COVID-19 cytokine storm surrogate marker:D-dimer | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker:D-dimer
Changes from baseline of COVID-19 cytokine storm surrogate marker:platelets | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker:platelets
Changes from baseline of COVID-19 cytokine storm surrogate marker: triglycerides | from Day 2 and until the end of hospitalization, Day 29 as a maximum
  Changes from baseline of COVID-19 cytokine storm surrogate marker: triglycerides
The time period until National Early Warning Score 2 (NEWS2) ≤ 2 during 2 consequent days is reached | from Day 1 and until the end of hospitalization, Day 29 as a maximum
  The time period until National Early Warning Score 2 (NEWS2) ≤ 2 during 2 consequent days is reached
The time period until National Early Warning Score 2 (NEWS2) ≤ 4 during 2 consequent days is reached | from Day 1 and until the end of hospitalization, Day 29 as a maximum
  The time period until National Early Warning Score 2 (NEWS2) ≤ 4 during 2 consequent days is reached

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm